CLINICAL TRIAL: NCT04635787
Title: ICU-Grade Wearable Sensors With Novel Respiratory Biomarkers to Diagnose and Detect Pre- and Very Early Symptomatic COVID-19 Infection Using Predictive Machine Learning Algorithms
Brief Title: Vital Sensor Monitors for CV19 Detection
Status: Completed | Type: Observational
Sponsor: Northwestern University (Other)
Collaborators: United States Department of Defense (U.S. Federal Agency)
Responsible Party: Principal Investigator, Shuai (Steve) Xu, Principal Investigator, Northwestern University
Other Study IDs: STU00213040
Record Dates: First submitted 2020-11-13; First posted 2020-11-19 (Actual); Last update posted 2023-05-06 (Actual); Status verified 2023-05

CONDITIONS: Covid19
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Healthy Adults: Adults 18 years or older
  Interventions: Device: ANNE One
- COVID19: Adults 18 years or older diagnosed with COVID 19
  Interventions: Device: ANNE One

INTERVENTIONS:
Device: ANNE One — Wireless vital sign monitoring device

SUMMARY:
This study will monitor physical bio-markers such as heart rate, respiratory rate, and temperature to detect potential COVID-19 infections.

DETAILED DESCRIPTION:
The purpose of this research is to assess the accuracy of wearable sensors at detecting and monitoring COVID-19 infections. Our small, wearable sensor can get data on your respiration, body temperature, heart rate, and blood oxygen level, which may help physicians better identify if a respiratory condition is worsening overtime. If successful, our sensor could help healthcare professionals detect early symptoms of COVID-19 respiratory infection and monitor recovery and treat people before their condition worsens significantly.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 18 years old or over
* Recent (within 1 week) occupational or home exposure to a newly diagnosed COVID-19 infected individual
* Able and willing to give written consent and comply with study procedures

Exclusion Criteria:

* Inability to understand instructions and follow a three step command
* The subject is pregnant, nursing or planning a pregnancy
* Inability to provide written consent
* Past confirmed COVID-19 infection with resolution of symptoms
* Past confirmed COVID-19 active infection moderate or severe symptoms

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Healthy adults and adults exposed to or diagnosed with COVID19
Sampling Method: Non-Probability Sample
Enrollment: 324 (Actual)
Dates: Start 2020-11-05 (Actual); Primary Completion 2021-03-31 (Actual); Study Completion 2021-08-31 (Actual)

PRIMARY OUTCOMES:
1.Efficacy of wearable device to detect respiratory infection parameters: cough count | 1 year
  Device data measuring cough count. Captured by analysis of peak acclerometer graphing and duration in meters per second squared (m/s2).

SECONDARY OUTCOMES:
2.Monitoring of respiratory infection symptoms, WURSS-11 Survey | Time Frame: 1 year
  WURSS-11 survey. https://www.fammed.wisc.edu/files/webfm-uploads/documents/research/wurss-11.pdf The WURSS-11 survey will be conducted on a weekly basis by study subjects for the duration of the study (up to 52 weeks).

CONTACTS AND LOCATIONS:
Locations (1):
- Northwestern Memorial Hospital, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No